CLINICAL TRIAL: NCT05727605
Title: Neurocognition After Radiotherapy in Adult Brain and Base of Skull Tumors
Brief Title: Neurocognition After Radiotherapy in CNS- and Skull-base Tumors
Acronym: NARCiS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: University Hospital, Ghent (Other); Gasthuis Zusters Antwerpen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S65664
Record Dates: First submitted 2023-01-13; First posted 2023-02-14 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-04

CONDITIONS: Cognition; Brain Tumor; Magnetic Resonance Imaging; Meningioma; Glioma; Pituitary Adenoma
MeSH Terms: conditions — Brain Neoplasms; Meningioma; Glioma; Pituitary Neoplasms | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Primary brain and skull-base tumors (Other): Primary brain and skull-base tumors who are amenable for radiotherapy (photon or proton therapy) will all be examined with neurocognitive tests, questionnaires and advanced MR imaging
  Interventions: Behavioral: Neurocognitive tests: WAIS digit span, HVLT-R, COWAT, MOCA, WAIS digit symbol substitution, TMT A&B, Stroop Color Word Test; Diagnostic Test: MRI; Behavioral: Questionnaires: EORTC QLQ C30 & BN20, STAI, CFQ, BDI-II, BRIEF-A, FACIT-F, PSQI; Other: Toxicity scoring

INTERVENTIONS:
Behavioral: Neurocognitive tests: WAIS digit span, HVLT-R, COWAT, MOCA, WAIS digit symbol substitution, TMT A&B, Stroop Color Word Test — Primary brain tumour patients will be evaluated longitudinally at the following timepoints: baseline (minimal 4 weeks after surgery, before radiotherapy), three months after end of radiotherapy, 1 year after end of radiotherapy and 2 years after end of radiotherapy. At each visit, neurocognitive testing, a self-report inventory and/or advanced MR imaging will take place.
  Time points: baseline, 12 months post-radiotherapy and 24 months post-radiotherapy
Diagnostic Test: MRI — Advanced MRI: all participants will be scanned on a 3T Siemens of Philips MR scanner (multicenter protocol): MPRAGE, FLAIR, T2, DWI, rsfMRI, SWI & ASL
  Time points: baseline, 3 months post-radiotherapy and 12 months post-radiotherapy
Behavioral: Questionnaires: EORTC QLQ C30 & BN20, STAI, CFQ, BDI-II, BRIEF-A, FACIT-F, PSQI — Time points: baseline, 12 months post-radiotherapy and 24 months post-radiotherapy
Other: Toxicity scoring — During and after radiotherapy and at at the end of the study, adverse events will be monitored using CTCAEv5.0.

SUMMARY:
The goal of this multicenter prospective longitudinal study is to study the long-term impact of multimodal treatment (chemotherapy, radiotherapy and surgery) in adult brain and base of skull tumors on neurocognitive functioning.

All included patients will complete a self-report inventory (subjective cognitive functioning, QoL, confounders), a cognitive test battery, an advanced MR at multiple timepoints. Moreover, toxicity will be scored according to the CTCAEv5.0 in these patients over time.

DETAILED DESCRIPTION:
This study will combine MR imaging techniques together with elaborate neuropsychological assessments and RT dosimetry in 120 patients who will be examined baseline (before RT) and followed longitudinally after RT.

The first objective is to build an NTCP model for neurocognitive decline after RT (for each cognitive domain separately), linking dose-volume parameters to structures within the brain susceptible to neurological damage and neurocognitive decline after radiotherapy. These NTCP models can be used to make predictions on neurocognitive decline in future primary brain tumour patients receiving cranial RT.

The second objective is to evaluate dose-dependent neurocognitive decline. In particular, the investigators will assess:

* Prevalence and severity of neurocognitive decline after RT for all cognitive domains
* Brain structures or functional brain connections important in neurocognitive functioning (based on dedicated MRI).
* Dose-dependencies of specific neurocognitive skills after RT in adult brain tumour patients
* Correlations between RT dosimetry and early brain changes (MRI)

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years at the time of diagnosis) with a primary brain or base of skull tumour, who are amenable for conventionally fractionated radiotherapy (photon or proton irradiation)

Exclusion Criteria:

* Patients with tumours with poor prognostic characteristics:

  * Incompletely resected IDH-wild-type glioma
  * Completely resected IDH-wild-type and MGMT-promotor unmethylated glioma
  * grade III meningioma
  * H3K27M+ midline glioma
* Patients with tumours requiring craniospinal irradiation (CSI)/whole ventricular irradiation (WVI)
* Hypofractionated/stereotactic radiation (fraction sizes > 2 Gy per fraction)
* Inability to perform the cognitive tests or self-report inventories because of motor/sensory deficits or insufficient Dutch language proficiency
* Mental retardation documented before diagnosis
* Pre-diagnosis/pre-existing psychiatric diagnosis resulting in cognitive deficits like psychoses, neurodevelopmental disorders (autism/learning disorders)
* Relapse previously treated by chemo and/or radiation therapy
* Genetic syndrome (e.g. Down)
* Unable to perform MR imaging (claustrophobia, metallic implants like pacemaker/ICD/neurostimulator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-02-08 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of neurocognitive decline (changes in z-scores) compared to baseline at one year post-radiotherapy, for all cognitive domains (memory, executive functioning, attention and language) | 2 years
Development of a Normal Tissue Complication Probability model (NTCP-model) for each cognitive domain (memory, executive functioning, attention and language) | 4 years
  Construct NTCP models to predict neurocognitive decline based on RT dosimetric and other explanatory variables (gender, age at diagnosis, comorbidities, level of education, social factors such as social activity and occupation, tumour size and localization, pathological/genetic/molecular characteristics, therapy protocols (surgery, radiotherapy and/or chemotherapy)) in an NTCP model for each cognitive domain

SECONDARY OUTCOMES:
Early (3 months post-radiotherapy) changes identified on structural and functional MR imaging (graph measures) | 4 years
  Changes on advanced MR imaging at 3 months post-RT compared to baseline
Late (12 months post-radiotherapy) changes identified on structural and functional MR imaging (graph measures) | 4 years
  Changes on advanced MR imaging at 12 months post-RT compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Maarten Lambrecht, MD PhD, Principal Investigator — UZ Leuven
Locations (3):
- Belgium (3):
  - University Hospitals Ghent, Ghent
  - UZ Leuven, Leuven
  - Gasthuis Zusters Antwerpen, Wilrijk

IPD SHARING:
Plan to Share IPD: No